## Imperial College London

## Consent Form for Participants Able to Give Consent

## Centre name:

Study Protocol number: 24SM8819

Full Title of Project: Ankle Arterial Doppler Waveform Assessment For Surveillance

Following Lower Limb Revascularisation: WAVE- study

Name of Principal Investigator:

| | | _ | | _ | _ | |
|------|----|----|------|---|-----|---|
| وما | ~~ | in | itia | | has | , |
| פסוט | 22 | ın | ItIa | | hai | |

| vers<br>For<br>and<br>fully | |
|---|---|
| at a | derstand that my participation is voluntary, and I am free to withdraw ny time without giving any reason and without affecting my legal rights eatment/healthcare. |
| capa<br>and | ng the study, if my clinical care team determines that I have lost the acity to provide informed consent, I will be withdrawn from the study, any identifiable data collected with consent will be retained and used e study. |
| be lo<br>Coll | derstand that sections of any of my medical notes and study data may booked at by researchers from Imperial College London,Imperial ege Healthcare NHS Trust, regulatory authorities where it is relevant by taking part in this research |
| supp<br>med<br>com | e/do not give consent for information collected about me to be used to cort other research or in the development of a new test, medication, lical device or treatment by an academic institution or commercial pany in the future, including those outside of the United Kingdom ch Imperial has ensured will keep this information secure). |
| | e/do not give consent to inform my GP or other health/ care essional. |
| Coll-<br>inve | derstand that the data collected from me are a gift donated to Imperial ege. I will not personally benefit financially if this research leads to an ntion and/or the successful development of a new test, medication tment, product or service. |
| part | e/do not give consent to being contacted about the possibility to take in other research studies. |
| | nsent to take part in (Ankle Arterial Doppler Waveform Assessment Surveillance Following Lower Limb Revascularisation: WAVE study). |

| Name of participant | Signature | Date |
|---------------------|-----------|------|

## Imperial College London

| Name of person taking consent | Signature | Date |
|--------------------------------------------|-----------|------|
| (if different from Principal Investigator) | | |

1 copy for participant; 1 copy for Principal Investigator

To ensure confidence in the process and minimise risk of loss, all consent forms <u>must</u> be printed, presented and stored in double sided format